CLINICAL TRIAL: NCT00678990
Title: Open Study to Evaluate Safety and Efficacy of Allogenic Islet Transplantation Using Islets Coated With Immobilised Heparin
Brief Title: Heparinized Islets in Clinical Islet Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Corline Biomedical AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAL-01
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Islets of Langerhans; islets; heparin
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open, single arm (Experimental): Transplantation of islets with heparin coating.
  Interventions: Procedure: Transplantation of islets with heparin coating

INTERVENTIONS:
Procedure: Transplantation of islets with heparin coating — Transplantation of islets with heparin coating

SUMMARY:
In this study the islets will be surface modified to carry immobilised heparin (Corline Heparin Conjugate) prior to transplantation. The primary objective is to investigate safety and efficacy of allogeneic islet transplantation using islets coated with immobilised heparin. The modification with heparin has been shown to protect the islets from being attacked by the immediate defence systems in blood (coagulation and inflammation), so that a larger portion of the islets will survive the initial phase and engraft. Evaluation will be based on metabolic and blood chemistry parameters.

DETAILED DESCRIPTION:
Transplantation of islets of Langerhans isolated from donated organs is a promising therapy for diabetes type 1. The results so far have, however, not met with the expectations due to relatively low efficiency. Even in situations where the patients have become insulin-free, it has been estimated that the transplanted islet mass is less than 25% of the islet mass of a healthy individual, which in many cases has required repeated use of insulin injections. The islets are transferred to the patient by an infusion drop to the liver via the portal vein.

Researches within the Nordic Network for Clinical Islet Transplantation have in a series of publications shown that the islets are subject to a violent immunological reaction that is non-specific with regard to the individual patient (IBMIR) during the initial contact with blood (Moberg et al, Lancet 2002, among several). The IBMIR reaction is in the earliest phase mediated by coagulation and complement reactions.

In this study the islets will be surface modified to carry immobilised heparin (Corline Heparin Conjugate) prior to transplantation. The primary objective is to protect the islets from being attacked by IBMIR so that a larger portion of the islets will survive the initial phase and engraft. In a paper published by the research group (Cabric et. al., Diabetes, May 2007), the beneficial effects of immobilised heparin on the islets to counteract IBMIR were shown by experiments at the lab bench and in experimental animals.

The evaluation of the transplantations in this study will be based on metabolic and blood chemistry parameters, similar to the evaluations of other transplanted patients within the Nordic Network.

ELIGIBILITY:
Inclusion Criteria

1. Male and female patients age 18 to 65 years of age.
2. Ability to understand and provide written informed consent.
3. Mentally stable and able to comply with the procedures of the study protocol.
4. Clinical history compatible with type 1 diabetes with onset of disease at < 40 years of age and insulin-dependence for > 5 years at the time of enrolment.
5. Stimulated C-peptide < 0.3 ng/mL (0.1 nmol/L) in response to a MMTT, before first islet transplantation.
6. All subjects must have received medical treatment of their diabetes under the guidance from an experienced endocrinologist.

   If not previously transplanted the patient must also have;
7. At least one episode of severe hypoglycaemia in the past 1 year defined as an event with at least one of the following symptoms; memory loss, confusion, uncontrollable behaviour, unusual difficulty in awakening, suspected seizure, loss of consciousness, or visual symptoms, in which the subject was unable to treat him/herself and which was associated with either a blood/plasma glucose level < 54 mg/dl (3.0 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration OR
8. Reduced awareness of hypoglycaemia as defined by a Clarke score of 4 or more.

Exclusion Criteria

Patients who meet any of these criteria are not eligible for participation in the study:

1. Patients with prior organ transplants other than a kidney graft and/or islets.
2. Patients with body mass index (BMI) > 30.
3. Insulin requirement > 1 Unit/kg/day at screening.
4. Consistently abnormal liver function tests (> 1.5 x ULN on two consecutive measurements > 2 weeks apart), at screening.
5. Proliferative untreated diabetic retinopathy
6. Increased risk for thrombosis (ex. homozygous APC-resistance) or bleeding (INR>1.5)
7. Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin
8. Patients with increased cardiac risk defined as;

   1. unstable coronary artery disease requiring hospitalization or revascularization within 6 months prior to baseline visit
   2. chronic heart failure which required hospitalization 30 days prior to baseline visit
9. Patients with active infections, unless treatment is not judged necessary by the investigators
10. Patients with serological evidence of infection with HIV, hepatitis B (patients with serology consistent with previous vaccination and a history of vaccination are acceptable) or hepatitis C.
11. Patients with active peptic ulcer disease, symptomatic gallstones or portal hypertension.
12. Patients who are pregnant or breastfeeding, or who intend to become pregnant.
13. Sexually active females who are not:

    1. post-menopausal,
    2. surgically sterile, or
    3. using a highly effective method of contraception, such as: intra uterine device, oral contraceptives, implants, injectables or barrier devices combined with spermicidal gel
14. Active alcohol or substance abuse
15. Patients with evidence of high-level sensitization (PRA> 50% with flow cytometry).
16. Patients with psychological conditions that make it unsafe to undergo islet transplantation or which preclude compliance with prescribed therapy
17. HbA1c >11% (International standard) corresponding to IFCC calibration 97 mmol/mol, at screening.
18. Medical history of egg allergy
19. Patients with any condition or any circumstance that in the opinion of the investigator would make it unsafe to undergo an islet transplant
20. Patients participating in or having participated in any other clinical drug studies in the past four weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Safety | 105 days
  Number of and grade of Serious Adverse events during the first 105 days after transplantation and Adverse events during the first 75 days after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Lorant, Principal Investigator — Uppsala University Hospital
Locations (2):
- Sweden (2):
  - Department of Transplantation Surgery, Karolinska University Hospital, Stockholm
  - Department of Transplantation and Liver Surgery, Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No